CLINICAL TRIAL: NCT04132921
Title: Risk Factors Related to Postoperative Acute Kidney Injury in Elderly Patients Undergoing Joint Replacement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Jin Dong Liu, The Affiliated Hospital of Xuzhou Medical University, Xuzhou Medical University
Other Study IDs: XYFY2020-KL050-01
Record Dates: First submitted 2019-10-11; First posted 2019-10-21 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2019-10

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with AKI: Patients with AKI after joint replacement
- Patients without AKI: Patients without AKI after joint replacement

SUMMARY:
Total hip arthroplasty refers to the replacement of the femoral head and acetabulum damaged by disease or trauma with an artificial hip joint, thereby restoring joint activity and original function. Acute kidney injury is a common complication after total hip arthroplasty. Previous studies have shown that the incidence of acute kidney injury after hip replacement is as high as 21.9%. Acute kidney injury has become a global safety issue, and the occurrence of acute kidney injury can lead to an increase in hospital stay, medical costs and increased risk of death.There is currently no global survey of the incidence of AKI, and only a number of studies have been conducted on specific patient groups (eg, inpatients, intensive care units [ICU] patients or children) due to differences in study design and definition of acute kidney injury.

DETAILED DESCRIPTION:
The incidence and prevalence of different studies vary widely, ranging from 0.32% to 44.30%. There are few studies on the risk factors associated with acute kidney injury after total hip arthroplasty, and early acute kidney injury is often overlooked due to the limitations of the current KDIGO-based diagnostic method. Therefore, it is particularly important for clinicians to understand the risk factors for postoperative acute kidney injury .

ELIGIBILITY:
Inclusion Criteria:

* Patients age 65 or older
* One-sided joint replacement;
* ASA score grade I-III

Exclusion Criteria:

* Emergency surgery patients;
* Patients with severe liver and kidney dysfunction;
* Missing related data;
* Serious systemic diseases before surgery;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adult patients who had undergone joint replacement between January 2014 and October 2019 were included . Patients developed AKI were deemed as cases, and those without AKI were included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and outcome of AKI after joint replacement | Within 7 days after surgery
  AKI can be diagnosed if one of the following conditions is true: (1) Serum creatinine increases by ≥26.5 μmol/L (0.3 mg / dl) within 48 h; (2)Serum creatinine rises more than 1.5 times of the baseline value, and is significantly or presumably the above situation occurred within 7 days;

SECONDARY OUTCOMES:
Possible risk factors for AKI after joint replacement | 1 day before surgery
  Patient's age, gender, height, weight
Intraoperative fluid volume and infusion type | during sugery and within 7days after surgery
  Record the total amount of infusion and infusion type of during surgery
Hemodynamic changes | during sugery and within 7days after sugery
  Focus on the fluctuation of mean arterial pressure
Factors related to anesthesia | during sugery and within 7days after sugery
  Record the type and dose of anesthetic used in the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jin Dong Liu, M.S, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bjerregaard LS, Jorgensen CC, Kehlet H; Lundbeck Foundation Centre for Fast-Track Hip and Knee Replacement Collaborative Group. Serious renal and urological complications in fast-track primary total hip and knee arthroplasty; a detailed observational cohort study. Minerva Anestesiol. 2016 Mar 30. Online ahead of print. PMID 27028450
- [Result] Yang L, Xing G, Wang L, Wu Y, Li S, Xu G, He Q, Chen J, Chen M, Liu X, Zhu Z, Yang L, Lian X, Ding F, Li Y, Wang H, Wang J, Wang R, Mei C, Xu J, Li R, Cao J, Zhang L, Wang Y, Xu J, Bao B, Liu B, Chen H, Li S, Zha Y, Luo Q, Chen D, Shen Y, Liao Y, Zhang Z, Wang X, Zhang K, Liu L, Mao P, Guo C, Li J, Wang Z, Bai S, Shi S, Wang Y, Wang J, Liu Z, Wang F, Huang D, Wang S, Ge S, Shen Q, Zhang P, Wu L, Pan M, Zou X, Zhu P, Zhao J, Zhou M, Yang L, Hu W, Wang J, Liu B, Zhang T, Han J, Wen T, Zhao M, Wang H; ISN AKF 0by25 China Consortiums. Acute kidney injury in China: a cross-sectional survey. Lancet. 2015 Oct 10;386(10002):1465-71. doi: 10.1016/S0140-6736(15)00344-X. PMID 26466051
- [Result] Maheshwari K, Turan A, Mao G, Yang D, Niazi AK, Agarwal D, Sessler DI, Kurz A. The association of hypotension during non-cardiac surgery, before and after skin incision, with postoperative acute kidney injury: a retrospective cohort analysis. Anaesthesia. 2018 Oct;73(10):1223-1228. doi: 10.1111/anae.14416. Epub 2018 Aug 24. PMID 30144029
- [Result] Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, Kurz A. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2017 Jan;126(1):47-65. doi: 10.1097/ALN.0000000000001432. PMID 27792044
- [Result] Magder SA. The highs and lows of blood pressure: toward meaningful clinical targets in patients with shock. Crit Care Med. 2014 May;42(5):1241-51. doi: 10.1097/CCM.0000000000000324. PMID 24736333